CLINICAL TRIAL: NCT05049668
Title: Long-term Follow-up of Patients Participating in RACE: the Prospective Randomized Multicenter Study Comparing Horse Antithymocyte Globuline (hATG) + Cyclosporine A (CsA) With or Without Eltrombopag as Front-line Therapy for Severe Aplastic Anemia Patients
Brief Title: RACE 2: a Long Term Follow-up of Patients Participating in the RACE Trial
Acronym: RACE2
Status: Enrolling by invitation | Type: Observational
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: EBMT-RACE 2
Record Dates: First submitted 2021-09-13; First posted 2021-09-20 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Antilymphocyte Serum; eltrombopag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- RACE 1 patients: After exiting the RACE trial (NCT02099747) patient will be invited to participate in this study
  Interventions: Drug: ATGAM plus CsA with or without Eltrombopag

INTERVENTIONS:
Drug: ATGAM plus CsA with or without Eltrombopag — Standard treatment with or without Eltrombopag
  Other Names: hATG+CsA +/- Revolade

SUMMARY:
After exiting the RACE trial (NCT02099747) patients will be invited to participate in this long term follow-up study

DETAILED DESCRIPTION:
Patients will be followed up annually, according to standard of care.

All diagnostic and therapeutic intervention will be performed according to standard of care, at discretion of the treating physician. In particular, during the study no extra Peripheral blood or Bone Marrow sampling will be performed, in addition to routine sampling for morphology and karyotype surveillance.

Molecular analysis by Next Generation Sequencing (NGS) will also be collected if the centre is doing this on a routine basis.

No Investigational Medicinal Product (IMP) or Non-Investigational Medicinal Product (NIMP) will be given to the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject participated in the RACE trial (NCT02099747, EudraCT number: 2014-000363-40) during which patient received ATGAM, Cyclosporine A with or without Eltrombopag.
2. Subject has provided informed consent to participate in long-term data collection

Exclusion Criteria:

None

Age Groups: Child, Adult, Older Adult
Study Population: Patients who participated in the initial RACE 1 trial
Sampling Method: Non-Probability Sample
Enrollment: 197 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2033-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Failure Free Survival | 15 years
  Failure Free Survival, where treatment failure is defined as one or more of the following: death, relapse, malignant clonal evolution, need for further (e.g. transplant)

SECONDARY OUTCOMES:
Response Rate: number of patients who reach a hematological response | 15 years
  Response Rate
Overall Survival | 15 years
  Overall Survival
Cumulative incidence of relapse after response | 15 years
  Cumulative incidence of relapse after initial hematological response (complete or partial)
Cumulative incidence of clonal evolution | 15 years
  Cumulative incidence of clonal evolution: Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome (MDS) or karyotypic abnormalities qualifying for the diagnosis of MDS (see World Health Organization (WHO) 2016)
Cumulative incidence of clinical Paroxysmal nocturnal hemoglobinuria (PNH) | 15 years
  Cumulative incidence of clinical PNH (hemolysis and/or thromboembolism), and of need of anti-complement treatment
Cumulative incidence of Solid Tumors | 15 years
  Cumulative incidence of solid tumours
Number of patients who need a Human Stem Cell Transplantation (HSCT) | 15 years
  Need for HSCT
Number of patients who need additional IST | 15 years
  Need for additional intensive Imune Suppressive Therapy (IST) (e.g. ATG, alemtuzumab or cyclophosphamide-based, or any other lymphocyte-depleting agent)
Number of patients who need Maintenance IST (e.g. CsA beyond 2 years) | 15 years
  Need for maintenance intensive IST (e.g. CsA beyond 2 years)
Number of patients who need additional Eltrombopag (EPAG) | 15 years
  Need for additional EPAG
Number of patients who need any other approved Aplastic Anemia (AA) treatment | 15 years
  Need for any other approved Aplastic Anemia (AA) treatment
Monitoring of Clonal Hematopoiesis of Indetermined Potential (CHIP) | 15 years
  As tracked by somatic mutations in genes associated with myeloid disorders

CONTACTS AND LOCATIONS:
Overall Officials: Regis Peffault de Latour, Prof, MD, Principal Investigator — Hospital St. Louis, Paris, France; Antonio M Risitano, MD, PhD, Principal Investigator — Hospital Avellino, Napels, Italy
Locations (1):
- Hospital St. Louis, Paris, France

IPD SHARING:
Plan to Share IPD: No